CLINICAL TRIAL: NCT04649801
Title: Catheter Ablation for Atrial Fibrillation in patientS With End-sTage Heart Failure and Eligibility for Heart Transplantation (CASTLE-HTx)
Brief Title: Catheter Ablation for Atrial Fibrillation in patientS With End-sTage Heart Failure and Eligibility for Heart Transplantation
Acronym: CASTLE-HTx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDZ_ER002_CS
Record Dates: First submitted 2020-10-07; First posted 2020-12-02 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure; Atrial Fibrillation
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional (No Intervention)
- interventional (Active Comparator)
  Interventions: Procedure: Atrial fibrillation ablation

INTERVENTIONS:
Procedure: Atrial fibrillation ablation — Catheter ablation
  Arms: interventional

SUMMARY:
CASTLE-HTx will determine if AF ablation has beneficial effects on mortality in patients with end stage HF who are eligible for HTx

DETAILED DESCRIPTION:
CASTLE-HTx is a randomized evaluation of ablative treatment of AF in patients with severe left ventricular dysfunction who are candidates and eligible for HTx. The primary endpoint is the composite of all-cause mortality, worsening of HF requiring a high urgent transplantation or LVAD implantation. The secondary study endpoints are all-cause mortality, cardiovascular mortality, cerebrovascular accidents, worsening of HF requiring unplanned hospitalization, AF burden reduction, unplanned hospitalization due to cardiovascular reason, all-cause hospitalization, QoL, number of delivered implantable cardioverter-defibrillator (ICD) therapies, time to first ICD therapy, number of device-detected ventricular tachycardia/ventricular fibrillation episodes, LV function, exercise tolerance, and percentage of right ventricular pacing. Ventricular myocardial tissue will be obtained from patients who will undergo LVAD implantation or HTx to assess the effect of catheter ablation on human HF myocardium.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic paroxysmal or persistent AF (paroxysmal: ≥2 symptomatic or one documented AF episode lasting 30 seconds or more in the last 3 months; persistent: ≥1 documented episode in the last 3 months).
2. Eligible for heart transplantation due to end-stage heart failure
3. LV dysfunction with left ventricular ejection fraction ≤ 35% (measured in the last 6 weeks prior to enrollment).
4. NYHA class ≥ II.
5. Indication for ICD therapy due to primary prevention.
6. Dual chamber ICD with Home Monitoring capabilities already implanted.
7. The patient is willing and able to comply with the protocol and has provided written informed consent.
8. Sufficient GPRS-network coverage in the patient's area.
9. Age ≥ 18 years.

Exclusion Criteria:

1. Documented left atrial diameter > 6 cm (parasternal long-axis view)
2. Contraindication for chronic anticoagulation therapy or heparin
3. Previous left heart ablation procedure for atrial fibrillation
4. Acute coronary syndrome, cardiac surgery, angioplasty, or cerebrovascular accident within 2 months prior to enrollment
5. Untreated hypothyroidism or hyperthyroidism
6. Enrollment in another investigational drug or device study
7. Indication for cardiac resynchronization therapy
8. Woman currently pregnant, breastfeeding, or not using reliable contraceptive measures during fertility age
9. Mental or physical inability to participate in the study
10. Listed as "high urgent" for heart transplantation
11. Cardiac assist device implanted
12. Planned cardiovascular intervention
13. Life expectancy ≤ 12 month
14. Uncontrolled hypertension
15. Requirement for dialysis due to end-stage renal failure
16. Participation in another telemonitoring concept

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Mortality or transplantation | 24 months
  composite of all-cause mortality, worsening of HF requiring a high urgent transplantation or implantation of a ventricular assist device

CONTACTS AND LOCATIONS:
Locations (1):
- Herz- und Diabeteszentrum NRW, Ruhr-Universität Bochum, Bad Oeynhausen, Germany

REFERENCES:
- [Derived] Sohns C, Fox H, Marrouche NF, Crijns HJGM, Costard-Jaeckle A, Bergau L, Hindricks G, Dagres N, Sossalla S, Schramm R, Fink T, El Hamriti M, Moersdorf M, Sciacca V, Konietschke F, Rudolph V, Gummert J, Tijssen JGP, Sommer P; CASTLE HTx Investigators. Catheter Ablation in End-Stage Heart Failure with Atrial Fibrillation. N Engl J Med. 2023 Oct 12;389(15):1380-1389. doi: 10.1056/NEJMoa2306037. Epub 2023 Aug 27. PMID 37634135